CLINICAL TRIAL: NCT01308840
Title: Phase II Study of Gemcitabine, Oxaliplatin in Combination With Panitumumab in Kras/B-raf Wild-Type Unresectable or Metastatic Biliary Track and Gallbladder Cancer
Brief Title: Gemcitabine, Oxaliplatin and Panitumumab in Kras/B-raf Wild-Type Biliary Track and Gallbladder Cancer
Acronym: UGIH09067
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Aram Hezel, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UGIH09067
Record Dates: First submitted 2010-08-09; First posted 2011-03-04 (Estimated); Results first posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-07

CONDITIONS: Biliary Tract Cancer; Gallbladder Cancer
Keywords: Unresectable; metastatic; biliary tract; gallbladder cancer
MeSH Terms: conditions — Biliary Tract Neoplasms; Gallbladder Neoplasms; Neoplasm Metastasis | interventions — Panitumumab; Oxaliplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Panitumumab (Experimental): Panitumumab 6mg/kg on days 1 and 15 of every cycle (28 days); Gemcitabine 1000mg/m2 on days 1 and 15 of every cycle (28 days); Oxaliplatin 85mg/m2 on days 1 and 15 of every cycle (28 days)
  Interventions: Drug: Panitumumab; Drug: oxaliplatin; Drug: gemcitabine

INTERVENTIONS:
Drug: Panitumumab — Day 1 and 15 = 6 mg/kg IV
  Other Names: GEMOX-Panitumumab (GEMOX-P)
Drug: oxaliplatin — Days 1 and 15 = 85mg/m2 IV
Drug: gemcitabine — Days 1 and 15 = 1000 mg/m2 IV

SUMMARY:
The purpose of this study is to determine disease response of GEMOX-Panitumumab (GEMOX-P) in KRAS/ BRAF wild-type, Stage IV, biliary tract and gallbladder cancer patients who have previously not received chemotherapy. This study will also examine the potential toxicities, progression-free and overall survival in this population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic or unresectable Kras and Braf wild-type biliary tract adenocarcinoma (bile ducts, hepatic duct, cystic duct, common bile duct, ampulla of Vater or gallbladder adenocarcinoma).
* Screening for tumor Kras and Braf mutations requires formalin fixed paraffin embedded tumor blocks from core needle excisional biopsy.
* Participants must have measurable disease.
* No prior chemotherapy for biliary tract or gallbladder cancer. Prior chemoembolization or radiation to the liver allowed as long as measurable disease outside chemoembolization or radiation area and other baseline characteristics met and at least 4 weeks has lapsed since therapy. No prior gemcitabine or oxaliplatin or anti-EGFR therapies including panitumumab therapy allowed.
* Age minimum 18 years old.
* Life expectancy of greater than 3 months.
* ECOG performance status < 1
* Participants must have normal organ and marrow function as defined below:
* Leukocytes > 3,000/mcL Absolute neutrophil count > 1,500/mcL Platelets > 100,000/mcL hemoglobin > 9mg/dL Mg > 1.2 mEq/L total bilirubin < 2.5 mg/dL AST (SGOT)/ALT (SGPT) < 2.5 X institutional upper limit of normal (unless liver is involved with tumor, in which case the transaminases must be 5 x upper limits of normal), creatinine within normal institutional limits or creatinine clearance > 60 mL/min/1.73 m2 for subjects with creatinine levels about institutional normal
* Patients with concurrent malignancy may be included if disease is characterized by one of the following definitions: 1. Malignancy treated with curative intent and with no known active disease present for 3 years prior to randomization and felt to be at low risk for recurrence by the treating physician. 2. Adequately treated non-melanomatous skin cancer or lentigo maligna without evidence of disease. 3. Adequately treated cervical carcinoma in situ without evidence of disease. 4. Prostatic intraepithelial neoplasia without evidence of prostate cancer. 5. DCIS without evidence of breast cancer.
* Ability to understand and the willingness to sign a written informed consent document.
* Patients may have prior placement of stents or shunts to relieve biliary obstruction.

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Participants may not be receiving any other study agents.
* Participants with known brain metastases.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine, oxaliplatin or panitumumab.
* Patients with preexisting peripheral neuropathy of grade 2 or greater severity according to the Common Terminology Criteria of the NCI (version 3.0) are ineligible.
* Patients with biliary obstruction with inadequate drainage and total bilirubin > 2.5 mg/dL are ineligible.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements,
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan.
* Known positive test(s) for HIV, hepatitis C virus, acute or chronic active hepatitis B infection.
* Pregnant women are excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aram Hezel, MD, Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - Dana-Farber / Harvard Cancer Center, Boston, Massachusetts
  - University of Rochester Medical Center, Rochester, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38 participants were screened.
Pre-assignment Details: 5 subjects were not eligible to enroll. 2 participants did not receive the intervention.
Period: Overall Study
Arm/Group | Panitumumab
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Panitumumab
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 61 [36 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 31
Eastern Cooperative Oncology Group (ECOG) Performance status [Number; unit: participants] — ECOG describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability. It ranges from 0-5 with higher numbers indicating reduced ability to care for themself.
  participants
    0 | 10
    1 | 21
Extent of disease [Number; unit: participants]
  locally advanced | 2
  metastatic | 29
primary tumor site [Number; unit: participants]
  intrahepatic cholangiocarcinoma | 25
  gallbladder | 3
  extrahepatic cholantiocarcinoma | 3
metastases [Number; unit: participants]
  lymph nodes | 24
  lung | 8
  bone | 4
  omentum/peritoneal | 4
  adrenal | 3
  pelvic soft tissue | 1

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Response to GEMOX-Panitumumab (GEMOX-P) in Chemotherapy naïve KRAS/ BRAF Wild Type Stage IV Biliary Tract Cancer Using the Response Evaluation Criteria In Solid Tumors (RECIST) Criteria.
Description: Tumor measurement - same imaging modality used in pre-treatment evaluation - include radiological examination of all areas with affected disease. For pretreatment and at the end of cycle 2 CT scans (chest/abdomen/pelvis) will be used. For all subsequent cycles, CT of chest/abdomen/pelvis will be used every 8 weeks.
Time Frame: end of cycle 2 of treatment
Measure: Number; unit: participants
Arm/Group | Panitumumab
Number analyzed (Participants) | 31
participants
  complete response | 0
  partial response | 14
  stable disease | 14
  progressive disease | 3

2. Secondary Outcome: Median Progression Free Survival
Description: Progression-free survival was defined as the time from study enrollment to date of cancer progression or death, whichever occurred first. Progression was assessed using CT scans and the Response Evaluation Criteria In Solid Tumors criteria. Progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: time to cancer progression or death
Measure: Median (Full Range); unit: months
Arm/Group | Panitumumab
Number analyzed (Participants) | 31
months | 10.6 [4.8 to 24.2]

3. Secondary Outcome: Median Overall Survival
Description: Death from any cause was used.
Time Frame: enrollment until date of death
Measure: Median (Full Range); unit: months
Arm/Group | Panitumumab
Number analyzed (Participants) | 31
months | 20.3 [9.1 to 25.1]

4. Secondary Outcome: The Number of Participants Who Experience an Adverse Event
Description: Any adverse event continuing after the study completion and considered potentially related to study treatment will be followed until resolution, stabilization or initiation of treatment that confounds the ability to assess the event
Time Frame: baseline to study completion
Measure: Number; unit: participants
Arm/Group | Panitumumab
Number analyzed (Participants) | 31
participants | 31

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of treatment.
Arm/Group | Panitumumab
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 31/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab (N=31)
Anaemia (Blood and lymphatic system disorders) | 26
neutropenia (Blood and lymphatic system disorders) | 7
Leukopenia (Blood and lymphatic system disorders) | 19
Thrombocytopenia (Blood and lymphatic system disorders) | 24
Fatigue (General disorders) | 25
Nausea (Gastrointestinal disorders) | 23
abdominal pain (Gastrointestinal disorders) | 9
diarrhea (Gastrointestinal disorders) | 14
infection (Infections and infestations) | 4
neuropathy (Nervous system disorders) | 21
rash (Skin and subcutaneous tissue disorders) | 20
elevated alkaline phosphatase (Hepatobiliary disorders) | 20
Hypomagnesemia (Blood and lymphatic system disorders) | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes